CLINICAL TRIAL: NCT00253773
Title: Metabolic Effects of Chemical Interactions in Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ES12929 (completed); DK66008
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Oxidative Stress
Keywords: sulfer amino acids; redox status
MeSH Terms: interventions — Acetaminophen; Cysteine; Methionine

INTERVENTIONS:
Drug: acetominophen, sulfer amino acids; cysteine and methionine

SUMMARY:
This pilot study tests the feasibility of using GSH redox state and high resolution proton NMR spectroscopy (1H-NMR) to detect metabolic changes due to acetominophen and sulfur amino acid deficiency. Our central hypothesis is that the a 2-day sulfur amino acid deficiency will alter acetominophen metabolism, acetominophen will affect sulfur amino acid homeostasis, and the treatments together will alter the global metabolic profile, as measured by 1H-NMR spectroscopy.

DETAILED DESCRIPTION:
Most occupational exposures to toxic chemicals occur in the context of complex mixtures, often in combination with varied diet, prescription drug use and disease. In principle, information-rich metabolic analyses provide an approach to study toxicologic consequences of such complex chemical interactions by revealing metabolic perturbations before irreversible injury occurs. This pilot study tests the feasibility of using GSH redox state and high resolution proton NMR spectroscopy (1H-NMR) to detect metabolic changes due to chemical interactions. The proposed model involves interaction of chemical exposure (2 doses of acetaminophen, APAP, 15 mg/kg) and 2 days of sulfur amino acid- (SAA-) free diet. 30% of APAP metabolism occurs through pathways dependent upon SAA metabolites and up to 50% of the RDA for SAA is needed to metabolize 2 doses of APAP. Both treatments are without toxicity in humans and both affect GSH homeostasis, which will be assessed in vivo by plasma measurements. Inter-individual variation will be minimized with each individual being his/her own control. Environmental and dietary influences will be controlled in a clinical research unit. Aim 1 is to determine whether SAA-free diet and APAP independently perturb GSH redox homeostasis. Aim 2 is to determine whether APAP intake interacts with SAA-free diet in affecting GSH redox state. Aim 3 is to use 1H-NMR spectroscopy to determine whether exposure to APAP and SAA-free diet interact in their effects on metabolic profile. The results will provide key data on the suitability and sensitivity of redox measurements and 1H-NMR spectroscopy for study of chemical interactions. This could provide a foundation for the use of perturbation of metabolic profile as a means to identify risks and consequences of complex chemical mixtures which would be especially relevant to occupational exposures in combination with therapeutic drugs and other health risk factors.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers males and females

Exclusion Criteria:

acute/chronic illnesses age less than 18 and greater than 40 pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
individual thiol and disulfide components; GSH/GSSG and Cys/CySS redox state; urinary output of taurine and sulfate

CONTACTS AND LOCATIONS:
Overall Officials: Dean Jones, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States